CLINICAL TRIAL: NCT03613922
Title: Effects of Early Manual Therapy on Functional Outcomes After Volar Plating of Distal Radius Fractures: A Randomized Controlled Trial
Brief Title: Effects of Early Manual Therapy on Functional Outcomes After Volar Plating of Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Murat TOMRUK, PhD, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TomrukDRF
Record Dates: First submitted 2018-07-26; First posted 2018-08-03 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Distal Radius Fracture
Keywords: manual therapy; radius fracture; function; disability; physiotherapy
MeSH Terms: conditions — Wrist Fractures; Radius Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Manual Therapy Group (Experimental): Routine physiotherapy program plus Mulligan's Mobilization with Movement technique were applied.
  Interventions: Other: Early Manual Therapy; Other: Routine Physiotherapy
- Routine Physiotherapy Group (Active Comparator): Only routine physiotherapy program was applied
  Interventions: Other: Routine Physiotherapy

INTERVENTIONS:
Other: Early Manual Therapy — Mulligan's Mobilization with Movement technique for radiocarpal,ulnocarpal, distal radioulnar and proximal radioulnar joints was applied.
  Arms: Early Manual Therapy Group
Other: Routine Physiotherapy — Routine physiotherapy program consisted of range of motion, flexibility and strengthening exercises, and home exercise program was applied.

SUMMARY:
The aim of the study was to investigate the effects of early manual therapy on function, pain, range of motion (ROM), hand and pinch grip strength and disability level in patients underwent volar plating after distal radius fracture (DRF). Patients were randomly divided into two groups: Routin Physiotherapy (RP) or Early Manual Therapy (EMT). While RP group received routine physiotherapy, EMT group received routine physiotherapy plus Mulligan's Mobilization With Movement technique. All treatments were done two sessions a week, through 12 weeks. Function, pain, range of motion (ROM), hand and pinch grip strength and disability level of patients were assessed. Measurements were made at postoperative week 3, 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* An age of eighteen years or older
* An unstable fracture of the distal end of the radius
* Fixation with a volar locking plate
* Able to read, write, and understand Turkish
* Willing and able to attend the study

Exclusion Criteria:

* Previous fracture on the injured side
* Concurrent fracture in contralateral upper extremity
* Accompanied bony and soft tissue injuries other than radius fracture
* Inflammatory joint diseases, metabolic diseases and neurological diseases
* Mental and cognitive disorders that would seriously affect cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
change in the function | postoperative week 6, 12.
  Function was asssesed by using Patient Rated Wrist Evaluation (PRWE)

SECONDARY OUTCOMES:
change in the severity of pain | postoperative day 1, postoperative week 3, 6, 12.
  Severity of pain was assessed by using Visual Analogue Scale (VAS), which ranges between 0-10 points, 0 represents no pain and 10 denotes maximum pain intensity.
change in the range of motion (ROM) | postoperative week 3, 6, 12.
  ROM was assesed by using an universal goniometer
change in hand and pinch grip strength | postoperative week 3, 6, 12.
  hand and pinch grip strength was assesed by using hydrolic hand and finger dynamometers.
change in disability | postoperative week 6, 12.
  Disability level was assesed by using Disabilities of Arm, Shoulder and Hand (DASH) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No